CLINICAL TRIAL: NCT06615037
Title: Isokinetic Strength Profile of Hip Joint in Females With Primary Dysmenorrhea During Different Phases of Menstrual Cycle
Brief Title: Strength Profile of Hip Joint in Females With Primary Dysmenorrhea During Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Mohamed Mitwally Amer, Principle Investigator, Cairo University
Other Study IDs: P.T.REC\012\005318
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; primary dysmenorrhea; Hip joint strength; isokinetic strength profile
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Symptomatic dysmenorrhea: According to WaLLID Scale Questionnaire
  Interventions: Other: Assess Hip joint strength by Biodex isokinetic dynamometer (System 4 Pro)
- Group B: Asymptomatic dysmenorrhea: According to WaLLID Scale Questionnaire
  Interventions: Other: Assess Hip joint strength by Biodex isokinetic dynamometer (System 4 Pro)

INTERVENTIONS:
Other: Assess Hip joint strength by Biodex isokinetic dynamometer (System 4 Pro) — Assessment of the strength of hip flexors and extensors muscles:
  * Participants will be in a supine-lying position, the highest reliability (ICC = 0.90) according to the results of the meta-analysis (Contreras et al., 2021).
  * Seat orientation 0°.
  * Dynamometer tilt 0° and orientation 0°.
  * The axis of the dynamometer on the greater trochanter of the femur.
  * The test parameters included a 0-90 degree range of motion.
  * During the isokinetic testing movement, the hip was first flexed from a neutral (starting) position to 90° (for hip flexion) and then the direction of the movement was reversed (for hip extension)
  * Angular speed at 120°/s which shows excellent reliability (ICC = 95%) with concentric contraction mode (Contreras et al., 2021) .

SUMMARY:
The goal of this observational study is to investigate the effect of primary dysmenorrhea on strength of hip joint muscles in females.

DETAILED DESCRIPTION:
The menstrual cycle is a physiological process in females manifested as periodic vaginal bleeding due to the shedding of the uterine lining (menstruation). Characterized by dynamic fluctuations in serum concentrations of several female sex steroid hormones. Estrogen, progesterone, follicle-stimulating hormone (FSH), and luteinizing hormone (LH) play a critical role in regulating the precise timing and events of the ovulatory cycle. Dysmenorrhea is considered a menstrual disorder and defined as painful menstrual cramps of uterine origin. It is classified as either primary or secondary dysmenorrhea (SD). Primary dysmenorrhea (PD) constitutes a prevalent gynecological condition in the absence of any identifiable pelvic pathology, characterized by cramping and severe pain localized within the lower abdomen. The prevalence of primary dysmenorrhea in females of reproductive age ranges from 45.0% to 94.0% in countries worldwide with 2% to 29% experiencing severe pain. A greater prevalence (70% to 90%) was generally reported among younger women (<24 years). Moderate and severe dysmenorrhea has even become a major reason for absenteeism from academic and professional settings and physical activity limitation in young women. Physical activity from standing, walking and balance to high impact sports was found to be directly influenced by the strength, power, and endurance of lower limb (LL) muscles especially hip muscles. Previous studies showed that the strength of LL muscles is influenced by the hormonal fluctuation that occurs during menstrual cycle phases.

These trial participants; will be divided into two groups:

(Group A): Female with symptomatic PD according to WaLLID scale. (Group B): Female with asymptomatic PD according to WaLLID scale.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 20 to 25 years.
* BMI ranges from 20 to 25 kg/m2.
* Having a regular menstrual cycle (28 ± 7 days with no intermittent bleeding).
* No pathology related to the pelvis.
* Having no injury in the lower limb.
* Not consuming contraceptives, dietary supplements and steroid drugs.

Exclusion Criteria:

* Menstrual irregularity.
* Pregnancy or suspicion of pregnancy.
* Having given birth.
* Using an intrauterine device.
* Oral contraceptives or antidepressant use.
* Having a diagnosis of secondary dysmenorrhea.
* Surgical history involving the abdominal region, pelvic region, and/or the spine in the last year.
* Having musculoskeletal problems related to lower extremities.
* Having any psychiatric or gynecological problems.
* Suffering from premenstrual syndrome.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult females Having a regular menstrual cycle (28 ± 7 days with no intermittent bleeding), No pathology related to the pelvis, Having no injury in the lower limb and Not consuming contraceptives, dietary supplements and steroid drugs.
Study Population: 44 adult females , age range: 20-25 years , BMI: 18-25 , 22 participants have symptomatic primary dysmenorrhea and 22 have asymptomatic primary dysmenorrhea according WaLLID Questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
1- Hip flexors isokinetic strength 2- Hip extensors isokinetic strength | 3 months
  The Biodex isokinetic dynamometer (System 4 pro) will be used to assess the strength of hip flexors and extensors during different phases of menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan Mohamed Mitwally Amer, Principal Investigator — Bachelor Physical Therapy- MUST; Amal Mohamed Yousef, Professor, Study Chair — Cairo University; Mai Mohamed Ali, Lecturer, Study Director — Cairo University; Ehab Kamal Mohamed Younis, lecturer, Study Director — Lecturer of obstetrics and gynecology - Faculty of Medicine - Misr university for science and technology
Locations (1):
- Cairo University, Giza, Egypt